CLINICAL TRIAL: NCT05613959
Title: Evaluation of the New Veress Needle+ Mechanism; A Study on Thiel-embalmed Bodies.
Brief Title: Evaluating the Novel Veress Plus Needle
Acronym: Veress+
Status: Completed | Type: Observational
Sponsor: Prof Jean Calleja-Agius (Other)
Responsible Party: Sponsor-Investigator, Prof Jean Calleja-Agius, Associate Professor; Head of Department of Anatomy, University of Malta
Organization: University of Malta (Other)
Other Study IDs: UM 0001
Record Dates: First submitted 2022-10-17; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Pneumoperitoneum
Keywords: Veress Needle; Thiel Embalmed Cadavers; Laparoscopy; Safety mechanism
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Veress +: The Veress+ system was used
  Interventions: Device: Veress +
- Veress conventional: The Conventional Veress needle was used
  Interventions: Device: Conventional Veress

INTERVENTIONS:
Device: Veress + — The Veress+ safety mechanism was used
  Groups: Veress +
Device: Conventional Veress — The Conventional Veress Needle was used
  Groups: Veress conventional

SUMMARY:
18 participants (novices, intermediates and experts) performed in total 248 insertions in a systematic way on Thiel embalmed bodies with wide and small bore versions of the conventional VNc (conventional Veress Needle) and the VN+(The Veress Needle plus). Insertion depth was measured by recording the graduations on the needle under direct laparoscopic vision.

DETAILED DESCRIPTION:
In total two Thiel embalmed bodies were used over three days. The first body was a 72 year old male with no previous laparotomy or abdominal scars, who had died of myocardial infarction (Length: 170 cm; bodyweight: 70 kg). The 2nd body was a male of 65 years without abdominal scars. The cause of death had been a hospital acquired pneumonia and pulmonary embolism secondary to metastatic pancreatic cancer (length186 cm; bodyweight: 80kg).

An Aesculap laparoscopy tower set up (Aesculap, 3773 Corporate Parkway, Center Valley, 18034 PA, USA) was used with a 10 mm 30 degrees scope, which was inserted through a balloon trocar (Medtronic Netherlands, Larixplein 4, 5616VB Eindhoven, The Netherlands) in the abdomen just below the umbilicus. Intra-abdominal pressure was stabilized using CO2 (Carbon Dioxide) to 4 mm Hg(Mercury). This pressure-level was as low as possible to allow for unambiguous visualization of the insertions but almost equalling normal abdominal pressure. Two different needle types were used, a thin bore needle with a diameter of 2 millimeter (mm) and a length of 145 mm and a wide bore with 2.8 mm diameter and 145 mm length. The study was registered under number FRECMDS-2021-134 of the Ethical Committee of Faculty of Medicine and Surgery of the University of Malta.

Questionnaire The investigators used a questionnaire which consisted of questions about gender, age and previous experience. A 1 to 5 Likert scale was used to score the "life-likeness" of the Thiel embalmed bodies, realism of the procedure, safety the VN+ procedure, and difficulty of using the new needle design.

Protocol After completing the first part of the questionnaire, the participants were instructed and explained how the mechanism works. During the instruction phase, they were allowed to try the needle on a dedicated area, away from the intended research area, until they were able to manage their grip and found their best insertion strategies. To minimize the risk of hitting organs upon entering the abdominal cavity, certain areas are dedicated for VN (Veress Needle) placement such as Palmer's point in the left upper quadrant of the abdomen. In order to use the bodies as efficiently as possible whilst offering a similar experience in terms of abdominal composition to all participants, the whole upper part of the abdomen was used for the insertions, which were done in an alternating fashion (with and without the safety mechanism) for 12 punctures (2x6) from cranial to caudal so a "fresh" part (with no defect or lesion) of abdominal wall was used for each attempt. The participants were with their backs to the video monitor so they were blinded to what was happening inside the abdomen. Insertion of the VN+ was successful when the mechanism fully unlocked. If not, the attempt was noted as an unsuccessful trial, the cause was determined and the insertion data was removed. After the hands- on part, the participants were asked to fill out the last part of the questionnaire with questions about the quality of the bodies and procedures based on their personal experiences and the difficulty of using the VN+ device. It is important to note that the VN+ dislodge action is not influenced by the amount of insertion force but only by the position of the inner stylet.

Data comparison and Statistical analysis Video footage was used by three observers to determine the insertion depth, indicated by the number of markings engraved on the part of the needle surface inside the abdomen. The true insertion depth was calculated in Excel based on the known distance between each marking. After the participants completed the tests, any differences in maximum insertion depth between the VNc and VN+ groups were determined with a Student's t-test (SPSS v16, SPSS, Inc., Chicago, IL). A p-value < 0.05 was considered a signiﬁcant difference. The same was done comparing the wide bore with the small bore needles and other variables including the different genders. The potential learning curve was established based on a regression analysis executed on the averaged outcomes per trial including all trial data. The potential influence of wear was established based on a regression analysis conducted on 12 separately executed trials with the wide bore needles. Wear is defined as diminishing sharpness of the bevel of the Veress needle after each attempt. For the regression analysis a p-value <0.05 was considered signiﬁcantly different.

ELIGIBILITY:
Inclusion Criteria:

* medical background, healthy

Exclusion Criteria:

* physically or mentally handicapped

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical residents, young surgeons, exeprienced surgeons from the University of Malta Mater Dei Hospital
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2021-09-26 (Actual)

PRIMARY OUTCOMES:
depth of insertion | 20 minutes
  the depth of insertion of the needle into the abdominal cavity

CONTACTS AND LOCATIONS:
Overall Officials: Jean Calleja Agius, MD PhD, Study Director — University of Malta
Locations (1):
- Laboratory for Anatomy, Valletta, Malta

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT05613959/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT05613959/ICF_001.pdf